CLINICAL TRIAL: NCT01599416
Title: Randomized, Double-blind, Placebo-controlled Study ,Oral U-relax in the Influence of the Vaginal Environment Health Promotion, and the HPV DNA Test Index Change From Positive to Negative on the HPV Infection Women
Brief Title: Influence of U-relax on Vaginal Health Promotion and HPV DNA Test Change From Positive to Negative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CGMH-O&G-201101TF01; 99-0948A3 (Other: CGMH)
Record Dates: First submitted 2012-05-07; First posted 2012-05-16 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2012-04

CONDITIONS: Human Papillomavirus; Vaginal Infection
Keywords: Oral Probiotics; HPV DNA Index Test; Vaginal infection
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Intervention Model Description: U-relax Group: U-relax capsules Day 1-5: take two capsuals of oral U-relax everyday before sleep Day 6-360: take one capsule of oral U-relax everyday before sleep
  Control Group: Placebo capsules Day 1-5: take two capsuals of oral placebo everyday before sleep Day 6-360: take one capsual of oral placebo everyday before sleep
Who Masked: Participant, Care Provider, Investigator
Masking Description: same capsule appearance and bottle without any marks for identification to participants, care providers and investigators except serial numbers
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- U-relax Group (Active Comparator): Day 1-5: take two capsuals of oral U-relax everyday before sleep Day 6-360: take one capsual of oral U-relax everyday before sleep
  Interventions: Dietary Supplement: U-relax
- Placebo Group (Placebo Comparator): Day 1-5: take two capsuals of oral placebo everyday before sleep Day 6-360: take one capsual of oral placebo everyday before sleep
  Interventions: Dietary Supplement: U-relax

INTERVENTIONS:
Dietary Supplement: U-relax — Oral U-relax Day 1-5: 2 capsuals before sleep Day 6-360: 1 capsual before sleep
  Other Names: GR-1 and RC-14

SUMMARY:
The purpose of this study is to understand the effect of using oral U-relax on HPV infected women for vaginal environment health promotion, and the HPV DNA Test Index change from positive to negative. Long-term infection of HPV is associated with cervical cancer. U-relax contains Lactobacillus GR-1 and Lactobacillus RC-14 and has been approved of its benefits on treatment of BV, UTI, IBD and can improve vaginal environment health. Patients with positive result of HPV DNA test have no appropriate and aggressive treatment to reduce the risk of cervical cancer. This clinical trial tries to reveal the influence of oral U-relax and patients with HPV DNA test positive result.

DETAILED DESCRIPTION:
This study is a prospective, double blind, randomized clinical trial. Vaginal health screening and HPV DNA Test are carried out from 80 patients with positive HPV DNA Test after conization for 6 months. All these patients will participant this study during the 360-day trial period. All health related conditions will be monitored at the same time.

ELIGIBILITY:
Inclusion Criteria:

* female
* age over 30
* PAP Test with NEGATIVE FOR INTRAEPITHELIAL LESION OR MALIGNANCY result
* HPV DNA Index Test with POSITIVE result after conization for 6 months
* not pregnant

Exclusion Criteria:

* cervical intraepithelial neoplasia before conization
* cervical cancer patient
* with GI surgery
* GI dysfunction
* need for long-term antibiotics treatment

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Vaginal environment health check | up to Day 360
  PAP Test, general check and health condition questionnaire

SECONDARY OUTCOMES:
HPV DNA Index Test Change | Day 1, Day 360
  HPV DNA Index Test, Health Condition Check

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Che Ou, MD, Study Director — CGMH; Hao Lin, MD, Principal Investigator — CGMH
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Ou YC, Fu HC, Tseng CW, Wu CH, Tsai CC, Lin H. The influence of probiotics on genital high-risk human papilloma virus clearance and quality of cervical smear: a randomized placebo-controlled trial. BMC Womens Health. 2019 Jul 24;19(1):103. doi: 10.1186/s12905-019-0798-y. PMID 31340789